CLINICAL TRIAL: NCT00323310
Title: A Phase III Multi-Center Open Label Study to Evaluate Safety and Efficacy of MultiHance at the Dose of 0.10 mmol/kg in Magnetic Resonance Imaging of the Central Nervous System in Pediatric Patients
Brief Title: Safety and Efficacy of MultiHance in Pediatric Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Adequate statistical power at 92 dosed pts to meet study objectives.
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Gianpaolo Pirovano, Executive Director, Corporate Medical Development, Bracco Diagnostics, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MH 110
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Central Nervous System Diseases
Keywords: disease of the central nervous system (brain or spine)
MeSH Terms: conditions — Central Nervous System Diseases | interventions — gadobenic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadobenate Dimeglumine (Experimental)
  Interventions: Drug: gadobenate dimeglumine

INTERVENTIONS:
Drug: gadobenate dimeglumine — A dose of 0.10 mmol/kg (i.e., 0.2 mL/kg) of 0.5 molar MultiHance was injected intravenously at a rate of 2 mL/sec as a single dose.
  Other Names: MultiHance

SUMMARY:
The purpose of this study was to assess the safety and enhancing properties of the magnetic resonance imaging (MRI) contrast agent MultiHance in children aged 2 to 17 years having central nervous system (CNS) disorders.

ELIGIBILITY:
Inclusion Criteria:

* Between 2 and 17 years of age
* Informed consent from parents
* Assent from patient where required
* Known or highly suspected disease of the CNS and referred for either cranial or spinal MRI examination

Exclusion Criteria:

* Contraindication to MRI
* Undergoing MRI in an emergency situation
* Known allergy to one or more of the ingredients in MultiHance
* Sickle cell anemia moderate to severe renal impairment
* Received another investigational compound within 30 days
* Pregnancy
* Lactating females
* Likely to undergo an invasive procedure within 72 hours of receiving MultiHance

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from April 2006 to July 2008 at 17 investigational sites. The blinded read was conducted from September 12, 2008 to September 26, 2008.
Pre-assignment Details: 94 patients enrolled; 92 patients dosed.
Groups:
- Gadobenate Dimeglumine: Contrast Agent, 0.10 mmol/kg injection
Period: Overall Study
Arm/Group | Gadobenate Dimeglumine
Started | 92
Completed | 89
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — a parent refused blood draw | 1
Not completed — did not complete the 24-hr f-up visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.59 (4.017)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 45
Region of Enrollment [Number; unit: participants]
  United States | 35
  Europe | 47
  Canada | 1
  China | 9

OUTCOME MEASURES:

1. Primary Outcome: Delineation of Lesion Border (Change From Pre to Pre+Postdose) for Reader 1
Description: 5-point scale (0=no delineation of lesion borders [lesion not identified in image, lesion borders not visible]; 1=poor border delineation [all borders poorly distinct, lesion not separated from surrounding tissues/structures/edema]; 2=moderate border delineation [border delineation fair/not complete, lesion not clearly separated]; 3=good border delineation [border delineation complete, lesion adequately separated]; 4=excellent border delineation [borders sharply/clearly distinct, lesion sharply separated]) paired assessment to compare the difference between pre to pre+postdose
Time Frame: pre-dose and immediately postdose
Population: Include all ITT population. The number of units analyzed are the total number of lesions assessed by the reader from the total number of participants.
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 148
Units on a Scale (0 to 4)
  Predose | 1.7 (1.16)
  Pre+Postdose | 3.0 (1.20)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [1.1 to 1.5], Standard Deviation 1.46

2. Primary Outcome: Delineation of Lesion Border (Change From Pre to Pre+Postdose) for Reader 2
Description: as for outcome 1
Time Frame: pre-dose and immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 135
Units on a Scale (0 to 4)
  Predose | 1.9 (1.15)
  Pre+Postdose | 3.1 (1.11)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.9 to 1.4], Standard Deviation 1.45

3. Primary Outcome: Delineation of Lesion Border (Change From Pre to Pre+Postdose) for Reader 3
Description: as for outcome 1
Time Frame: pre-dose and immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 131
Units on a Scale (0 to 4)
  Predose | 1.7 (1.19)
  Pre+Postdose | 2.4 (1.12)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.4 to 0.9], Standard Deviation 1.42

4. Primary Outcome: Visualization of Lesion Internal Morphology (Change From Pre to Pre+Postdose) for Reader 1
Description: 5-point scale (0=no visualization of lesion internal morphology (LIM) [lesion not identified in image, not visible]; 1=poor visualization of LIM [insufficiently depicted, intralesional features poorly identified]; 2=moderate visualization of LIM [not completely depicted, some intralesional features visible]; 3=good visualization of LIM [completely depicted, intralesional features adequately identified]; 4=excellent visualization of LIM [optimally depicted, intralesional features clearly identified and characterized]) paired assessment to compare the difference between pre to pre+postdose
Time Frame: pre-dose to immediately post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 148
Units on a Scale (0 to 4)
  Predose | 1.9 (1.18)
  Pre+Postdose | 3.2 (1.19)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [1.1 to 1.6], Standard Deviation 1.56

5. Primary Outcome: Visualization of Lesion Internal Morphology (Change From Pre to Pre+Postdose) for Reader 2
Description: as for outcome 4
Time Frame: pre-dose to immediately post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 135
Units on a Scale (0 to 4)
  Predose | 2.1 (1.17)
  Pre+Postdose | 3.2 (1.13)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.8 to 1.4], Standard Deviation 1.49

6. Primary Outcome: Visualization of Lesion Internal Morphology (Change From Pre to Pre+Postdose) for Reader 3
Description: as for outcome 4
Time Frame: pre-dose to immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 131
Units on a Scale (0 to 4)
  Predose | 1.4 (1.06)
  Pre+Postdose | 2.0 (1.23)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.4 to 0.8], Standard Deviation 1.20

7. Primary Outcome: Lesion Contrast Enhancement (CE) (Change From Pre to Pre+Postdose) for Reader 1
Description: 5-point scale (0=no lesion CE [lesion not identified in image, no contrast between lesion and surrounding normal brain/spine tissue]; 1=poor lesion CE [diff. in signal intensity (SI) poor, lesion barely identified, not possible to evaluate/measure size]; 2=moderate lesion CE [diff. in SI fair, lesion identified, not possible to evaluate/measure size]; 3=good lesion CE [diff. in SI adequate, lesion identified, size evaluated/measured]; 4=excellent lesion CE [diff. in SI marked, lesion identified, size measured]) paired assessment to compare the diff. between pre to pre+postdose
Time Frame: pre-dose and immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 148
Units on a Scale (0 to 4)
  Predose | 1.8 (1.16)
  Pre+Postdose | 3.0 (1.19)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [1.0 to 1.5], Standard Deviation 1.57

8. Primary Outcome: Lesion Contrast Enhancement (CE) (Change From Pre to Pre+Postdose) for Reader 2
Description: as for outcome 7
Time Frame: pre-dose to immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 135
Units on a Scale (0 to 4)
  Predose | 2.0 (1.20)
  Pre+Postdose | 3.2 (1.12)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.9 to 1.4], Standard Deviation 1.49

9. Primary Outcome: Lesion Contrast Enhancement (CE) (Change From Pre to Pre+Postdose) for Reader 3
Description: as for outcome 7
Time Frame: pre-dose to immediately postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale (0 to 4)
Units Other Than Participants: Lesions
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Number analyzed (Lesions) | 131
Units on a Scale (0 to 4)
  Predose | 1.4 (0.96)
  Pre+Postdose | 2.2 (1.41)
Statistical Analysis 1: Comparison: Gadobenate Dimeglumine; Paired t-test to compare change from pre to pre+postdose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — H0: udiff = 0; Ha: udiff not = 0; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [0.6 to 1.1], Standard Deviation 1.54

10. Primary Outcome: The Number of Patients Administered MultiHance (Gadobenate Dimeglumine) Reporting Adverse Events
Time Frame: up to 72 hours post dose
Population: Included all dosed patients (safety population).
Measure: Number; unit: Participants
Arm/Group | Gadobenate Dimeglumine
Number analyzed (Participants) | 92
Participants | 8

ADVERSE EVENTS:
Arm/Group | Gadobenate Dimeglumine
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 8/92
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobenate Dimeglumine (N=92)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be presented during scientific symposia or published in a scientific journal only after review by Bracco in accordance with the guidelines set forth in the applicable publication or financial agreement.